CLINICAL TRIAL: NCT00296933
Title: Memory Functioning and Antidepressant Treatment: A Randomized Controlled Trial Comparing Escitalopram and Bupropion XL
Brief Title: Memory Functioning and Antidepressant Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: GlaxoSmithKline (Industry); H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHN REB #05-0464-A
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Major Depression; Antidepressant; Pharmacotherapy; Memory functioning; Memory Impairment
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Memory Disorders | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram
Drug: Bupropion XL

SUMMARY:
Major Depressive Disorder (MDD) is a serious illness associated with considerable morbidity, risk of suicide and adverse social consequences (Montgomery et al., 1994a). Cognitive impairment is one of the three major symptom areas of MDD. Specifically, memory impairment and concerns are one of the most commonly reported complaints in MDD. While antidepressant (AD) treatments vary a great deal in their propensity to cause cognitive impairment, there remains a paucity of empirical evidence on the effects of AD treatment on neuropsychological indices of memory functioning in non-geriatric depressed individuals. Hence, comparative effects of various AD drugs on memory functioning remain unclear.The aim of this study is to evaluate multiple aspects of memory functioning (short-term, working memory, verbal, non-verbal, spatial and prospective memory) of MDD patients before and after 8 weeks of antidepressant treatment with bupropion XL or escitalopram.

DETAILED DESCRIPTION:
Purpose of the Present Study:

The purpose of the present study is to comprehensively evaluate memory functioning of MDD patients before and after 8 weeks of antidepressant treatment with bupropion-XL or escitalopram. A neuropsychological test battery will incorporate multiple aspects of memory functioning including: short-term & working memory; verbal, non-verbal, spatial and prospective memory.

Major Research Questions:

1. Which subtypes of memory at baseline are more impaired?
2. What is the relationship between memory impairment and symptom severity and previous number of episodes or duration of illness?
3. Is successful AD treatment associated with improvement in memory functioning?
4. Is there a main effect by AD type?
5. On which subtypes of memory do patients improve, worsen, or remain neutral in the 2 different AD groups? (Main effect of memory type?)
6. What is the relationship between change in memory function and symptomatic outcome?

Study Design:

This is a randomized, double-blind, double-dummy trial comparing the memory functioning of depressed subjects before and after 8 weeks of treatment with bupropion-XL as compared to escitalopram.

All consenting, eligible subjects will receive either active bupropion-XL or active escitalopram following the baseline visit. Doses will be fixed with an opportunity for dose reduction if subjects are unable to tolerate fixed dose.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age: 18-50
* Recurrent Major Depressive Disorder; current Major Depressive Episode with at least one prior episode
* HAM-D >16
* Able to give written informed consent
* Agree to use a reliable means of birth control during the study, as determined by the investigator (females of child-bearing potential only)

Exclusion Criteria:

* History of head injury or loss of consciousness for longer than 30 minutes
* Presence of primary anxiety disorder, bipolar I or II disorder, or psychotic disorders
* Presence of anorexia nervosa or bulimia nervosa
* Presence or history of epilepsy or other seizure disorders
* Presence of significant Axis II disorder based on investigator judgment
* Presence of significant unstable medical condition
* Presence or past history of ADHD or significant learning disability
* ECTs (unilateral) within the past 12 months or bilateral ECT (ever)
* More than 2 failed adequate antidepressant treatments in the current episode
* Pregnant or breast-feeding females
* Have received treatment within the last 30 days with an investigational drug
* Prior non-response to either bupropion-XL or escitalopram
* Current treatment with Zyban (bupropion hydrochloride)
* Antidepressant treatment within the last week (within the last 3 weeks fluoxetine)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-12

PRIMARY OUTCOMES:
General Verbal Memory-California Verbal Learning Test® -2nd ed (CVLT® -II)

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression - 17-Item
Clinical Global Impression Severity and Improvement Ratings
Short Term & Working Memory: Wechsler Memory Scales III
Nonverbal Memory - Faces
WMS III Logical Memory (Prose Recall)
Nonverbal Memory - Spatial Memory
Shipley Institute of Living Scale
Prospective Memory

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H Kennedy, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada